CLINICAL TRIAL: NCT02175992
Title: Quality of Life After Surgery for Pancreatic Carcinoma
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Prof. dr. I.Q. Molenaar, MD, PhD, Dr., UMC Utrecht
Other Study IDs: 13/546
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Patients Suspected for a Pancreatic (Pre-)Malignancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Pancreatic cancer has a high mortality rate. Patients with an intended curative resection show a median survival of 17-23 months. Therefore, quality of life is very important in this patient group. In this study, the effect of pancreatic surgery on quality of life is measured.

ELIGIBILITY:
Inclusion Criteria:

* patients with a suspected pancreatic malignancy
* eligible for surgery with curative intent
* being able to complete questionnaires in Dutch
* age >=18 years

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a suspected pancreatic malignancy
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-03; Primary Completion 2016-12-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 2 years
  To assess the influence of pancreatic surgery for patients with a pancreatic malignancy on health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Quintus Molenaar, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Department of Surgery, University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Heerkens HD, van Berkel L, Tseng DSJ, Monninkhof EM, van Santvoort HC, Hagendoorn J, Borel Rinkes IHM, Lips IM, Intven M, Molenaar IQ. Long-term health-related quality of life after pancreatic resection for malignancy in patients with and without severe postoperative complications. HPB (Oxford). 2018 Feb;20(2):188-195. doi: 10.1016/j.hpb.2017.09.003. Epub 2017 Oct 29. PMID 29092792